CLINICAL TRIAL: NCT02235324
Title: Phase II Study of Ziv-Aflibercept Followed by the Addition of 5-FU in the Third Line Setting of Metastatic Colorectal Cancer
Brief Title: Ziv-Aflibercept Followed by Ziv-Aflibercept, Fluorouracil, and Leucovorin Calcium in Treating Patients With Stage IV Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3C-13-7; NCI-2014-01806 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-14-00081; 3C-13-7 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Mucinous Adenocarcinoma of the Colon; Mucinous Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Signet Ring Adenocarcinoma of the Colon; Signet Ring Adenocarcinoma of the Rectum; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — aflibercept; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ziv-aflibercept, leucovorin calcium, fluorouracil) (Experimental): PHASE I:
  Patients receive ziv-aflibercept IV over 1 hour on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. At the time of progression, patients proceed to Phase II.
  PHASE II:
  Patients receive ziv-aflibercept IV over 1 hour, leucovorin calcium IV over 1 minute, and fluorouracil IV over 46 hours on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: ziv-aflibercept; Drug: leucovorin calcium; Drug: fluorouracil; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: ziv-aflibercept — Given IV
  Other Names: aflibercept; vascular endothelial growth factor trap; VEGF Trap; Zaltrap
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how long it takes colorectal cancer resistant to standard treatment to grow while receiving treatment with ziv-aflibercept, and how well adding fluorouracil and leucovorin calcium to ziv-aflibercept works in treating patients with stage IV colorectal cancer after they progress on ziv-aflibercept alone. Ziv-aflibercept may stop the growth of colorectal cancer by blocking the formation of tumor blood vessels. Fluorouracil and leucovorin calcium are drugs used in chemotherapy. Fluorouracil works to stop the growth of tumors cells by preventing the cells from growing and dividing. Leucovorin calcium helps fluorouracil work better. Adding fluorouracil and leucovorin calcium to ziv-aflibercept may be an effective treatment for patients who progress on ziv-aflibercept alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the progression-free survival during the first phase of the study (PFS1) in patients with metastatic colorectal cancer treated with single agent ziv-aflibercept after progressing on leucovorin calcium, fluorouracil, oxaliplatin (FOLFOX) and leucovorin calcium, fluorouracil, irinotecan hydrochloride (FOLFIRI) with bevacizumab +/- cetuximab or panitumumab.

II. To determine the progression-free survival (PFS2) in patients with metastatic colorectal cancer treated with ziv-aflibercept and 5-fluorouracil (fluorouracil), after progressing on ziv-aflibercept alone.

SECONDARY OBJECTIVES:

I. Overall survival. II. Response rate. III. Incidence and nature of adverse events. IV. Growth modulation index (ratio of PFS2/PFS1).

TERTIARY OBJECTIVES:

I. To determine relevant biomarkers which can distinguish patients with a progression free survival greater than 3 months on single agent ziv-aflibercept (tumor vascular endothelial growth factor [VEGF], vascular endothelial growth factor receptor [VEGFR]1 and 2, baseline plasma phosphatidylinositol glycan anchor biosynthesis, class F [PlGF]).

II. Plasma levels of VEGF-A, B, C, D, intercellular adhesion molecule 1 (ICAM), chemokine (C-X-C motif) ligand 1 (melanoma growth stimulating activity, alpha) (Gro alpha), hepatocyte growth factor (HGF), stem cell growth factor beta (SCGF beta) prior to treatment and with each cycle of therapy.

III. Single nucleotide polymorphisms (SNPs) of VEGFA, VEGFR1 & 2 & 3, interleukin (IL)8, angiopoietin-2 (Ang2), IL-6, ICAM, PlGF, neuropilin (NRP)1 & 2, chemokine (C-X-C motif) receptor 2 (CXCR2) and others in the angiogenic pathway.

IV. Tumor messenger ribonucleic acid (mRNA) expression levels of VEGF B, C, D, VEGFR 3; NRP 1, 2, and VEGF isoforms on biopsy specimens taken at trial initiation and upon disease progression and addition of 5-FU.

V. Correlation of biomarkers with toxicity of ziv-aflibercept alone and with 5-FU.

OUTLINE:

PHASE I: Patients receive ziv-aflibercept intravenously (IV) over 1 hour on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. At the time of progression, patients proceed to Phase II.

PHASE II: Patients receive ziv-aflibercept IV over 1 hour, leucovorin calcium IV over 1 minute, and fluorouracil IV over 46 hours on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV colorectal adenocarcinoma previously treated with FOLFOX and FOLFIRI and bevacizumab, receipt of cetuximab or panitumumab is not required, and has shown progression or intolerant of both oxaliplatin and irinotecan-based regimens; baseline tumor assessments must be done within 28 days of starting treatment
* Patients must have lesions that can be easily biopsied
* Representative tumor tissue specimens (paraffin block preferred)
* Signed informed consent prior to initiation of any study-specific procedure or treatment, including agreement to two biopsies during the study
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Able to comply with the protocol, including tissue and blood sampling
* Leukocytes >= 3,000 per mm^3
* Absolute neutrophil count >= 1,000 per mm^3
* Platelet count >= 75,000 per mm^3
* Hemoglobin >= 9 g/dL (may be transfused to maintain or exceed this level)
* Creatinine clearance according to the Cockcroft and Gault formula of >= 50 mL/min
* Urine for proteinuria should be < 2 +; patients discovered to have >= 2 + proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate < 1 g of protein in 24 hours
* Total bilirubin < 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase and alanine aminotransferase < 2.5 x ULN
* International normalized ratio =< 1.5 and activated prothrombin time =< 1.5 x ULN for patients not receiving anti-coagulation therapy
* The use of full-dose oral or parenteral anticoagulants is permitted as long as the international normalized ratio (INR) or activated partial thromboplastin time (aPTT) is within therapeutic limits (according to the medical standard of the enrolling institution), and the patient has been on a stable dose of anticoagulants for at least two weeks prior to the first study treatment
* Female patients should not be pregnant or breast-feeding

  * A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone hysterectomy or bilateral oophorectomy; OR
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e. has had menses at any time in the preceding 12 months)
  * Female patients with childbearing potential should agree to use effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) during the study and for a period of at least 6 months following the last administration of study drug
  * Female patients with an intact uterus (unless amenorrheic for the last 24 months) must have a negative serum pregnancy test within 7 days prior to randomization into the study
* Male patients must agree to use effective contraception during the study and for a period of at least 6 months following the last administration of study drugs, even if they have been surgically sterilized

Exclusion Criteria:

* Any prior systemic treatment with targeted antiangiogenic agents except for bevacizumab; receipt of cetuximab or panitumumab is not an exclusion criteria
* Radiotherapy to any site for any reason within 14 days prior to treatment
* Uncontrolled intercurrent illness including, but not limited to

  * Any of the following within 6 months prior to inclusion: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) class III or IV congestive heart failure, stroke or transient ischemic attack
  * Any of the following within 3 months prior to inclusion: grade 3-4 gastrointestinal bleeding/hemorrhage (unless due to resected tumor), treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism or other uncontrolled thromboembolic event
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in the study
* History of arterial thromboembolic events
* History of abdominal fistula formation, gastrointestinal perforation, or abdominal abscess within six months
* History or evidence of inherited bleeding diathesis or coagulopathy with a risk of bleeding
* Patients must not be pregnant or nursing
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study drug
* Any hemorrhage or bleeding event >= CTCAE grade 3 within 4 weeks prior to the start of study medication
* Non-healing wound, ulcer, or bone fracture
* Inadequately controlled hypertension (systolic blood pressure [SBP] > 150 mmHg, diastolic blood pressure [DBP] > 100 mg Hg)
* Known positivity for human immunodeficiency virus (HIV)
* Malignancies other than colorectal adenocarcinoma within 5 years prior to treatment, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, and ductal carcinoma in situ treated surgically with curative intent
* Clinically detectable (by physical exam) third-space fluid collections (e.g. ascites or pleural effusion) that cannot be controlled by drainage or other procedures prior to study entry
* Treatment with any other investigational agent, or participation in another investigational drug trial within 28 days prior to randomization
* Patients can withdraw consent anytime during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival during the first phase of the study | Period from the start of ziv-aflibercept to the date of radiographic or clinical progression, death, or within 30 days off treatment
  Point and precision estimates, median and its 95% confidence interval (CI) will be provided. To examine associations between biomarkers and PFS1, the difference in progression-free survival by each biomarker level will be detected.
Progression-free survival during the second phase of the study | Period from the start of fluorouracil with ziv-aflibercept to the date of radiographic or clinical progression, death, or within 30 days off treatment
  Using the Simon's 2-stage optimum design, there is a 90% power to detect improvement of adding fluorouracil to ziv-aflibercept on PFS2 and the type I error rate is 2.3%. Point and precision estimates, median and its 95% CI will be provided.

SECONDARY OUTCOMES:
Overall survival (OS) | Period from treatment initiation with single agent ziv-aflibercept to death, assessed up to 3 years
  OS will be summarized with Kaplan-Meyer plots to describe the outcome of patients treated on this protocol.
Response rate assessed using Response Evaluation Criteria in Solid Tumors 1.1 | Up to 3 years
  Response rates will be calculated as the percent of evaluable patients whose best response is a complete response or partial response, and exact 95% confidence intervals will be calculated for this estimate.
Incidence of adverse events graded according to NCI CTCAE version 4.0 | Within 30 days of the last administration of the study drug
  Toxicities observed at each leg of the study will be summarized in terms of type (organ affected, laboratory determination), severity (by NCI Common Toxicity Criteria and nadir or maximum values for the laboratory measures), time of onset, duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by leg and by course of therapy.

OTHER OUTCOMES:
Plasma levels of PIGF | Up to 3 years
  The association between each biomarker and PFS1 will be assessed by maximal x^2 square approach by identifying the optimal cut-off value for each biomarker and adjusting p value based on the bootstrap-like p values. The association between biomarkers and tumor response and OS will be analyzed using Fisher's exact and log-rank tests. Biomarker levels will be categorized based on optimal cutoff values determined in the analysis for PFS.
mRNA level of VEGFR1, VEGFR2, and VEGF-A | Up to 3 years
  The association between each biomarker and PFS1 will be assessed by maximal x^2 square approach by identifying the optimal cut-off value for each biomarker and adjusting p value based on the bootstrap-like p values. The association between biomarkers and tumor response and OS will be analyzed using Fisher's exact and log-rank tests. Biomarker levels will be categorized based on optimal cutoff values determined in the analysis for PFS.

CONTACTS AND LOCATIONS:
Overall Officials: Afsaneh Barzi, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States